CLINICAL TRIAL: NCT06546098
Title: Expanded Access to Inhaled Molgramostim Nebulizer Solution in Adults With Autoimmune Pulmonary Alveolar Proteinosis (aPAP)
Brief Title: Molgramostim Nebulizer Solution Expanded Access Program Protocol
Status: Available | Type: Expanded Access
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAV006-06
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
Keywords: surfactant accumulation; autoimmune; alveolar proteinosis; GM-CSF
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired; Pulmonary Alveolar Proteinosis | interventions — Colony-Stimulating Factors; regramostim

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Molgramostim nebulizer solution — Solution for inhalation
  Other Names: Recombinant human granulocyte-macrophage colony stimulating factor (rhGM-CSF)

SUMMARY:
Autoimmune pulmonary alveolar proteinosis (aPAP) is a rare disorder in which a material called surfactant builds up in the lungs and makes it hard to breathe. In addition to shortness of breath, people with aPAP can experience persistent cough, overwhelming fatigue, unintentional changes in weight, chest or back pain, suddenly feeling out of shape, and general discomfort.

Currently, there are no approved medications for aPAP in the United States, but the symptoms of aPAP can be treated with whole lung lavage (WLL). WLL is an invasive procedure that temporarily removes surfactant, and it can result in serious consequences like trauma to the lung, a collapsed lung, and prolonged requirement for artificial ventilation.

Savara is studying an investigational drug called molgramostim nebulizer solution to see if it activates the cells that help clear surfactant from the lungs, which improves oxygen transfer from the lungs to the bloodstream. Molgramostim nebulizer solution is administered by inhalation using a hand-held nebulizer. In clinical trials, molgramostim nebulizer solution has shown improvements in gas exchange and patient reported outcomes.

This expanded access program will make molgramostim nebulizer solution available to adult patients with diagnosed aPAP. Access must be obtained through the treating physician. Patients will dose molgramostim nebulizer solution 300 micrograms (mcg) once daily and be followed by their physician every 3 months to assess their clinical status and report any adverse events.

DETAILED DESCRIPTION:
Autoimmune pulmonary alveolar proteinosis (aPAP) is a rare disease mediated by autoantibodies targeting granulocyte macrophage colony-stimulating factor (GM-CSF), resulting in malfunctioning macrophages with impaired surfactant catabolism. The latter causes accumulation of surfactant in the alveoli, which has a negative impact on gas exchange between lung and blood. The clinical course of autoimmune PAP varies among patients with continuously slowly progressive disease in most patients, spontaneous improvement in a small percentage (5-7%), and rapid progression and/or pulmonary fibrosis, respiratory failure, and death in others. The most common cause of death is respiratory failure followed by secondary pulmonary bacterial infections. Estimated 5-year mortality rates vary between 10-30%, with overall disease-specific survival rates at 5 years exceeding 80%.

There are currently no approved pharmacological treatments for aPAP in most of the world. Whole lung lavage (WLL) is the primary treatment option currently available for most aPAP patients. However, its invasive nature, limited access, and the variable effect of WLLs due to lack of standardization emphasize that there is an unmet need for a non-invasive, safe and well-tolerated, easily accessible and effective treatment for aPAP patients.

The rationale for treating aPAP patients with molgramostim nebulizer solution is based on the capacity of GM-CSF to promote differentiation and mobilization of different myeloid leukocyte subsets including neutrophils, tissue macrophages/dendritic cells or their circulating precursors. It is crucially involved in anti-microbial pulmonary host defense and ameliorates lung injury by increasing the size and activation of the alveolar macrophage pool. GM-CSF also contributes to the proliferation of megakaryocytic and erythroid progenitors and plays a key role in surfactant homeostasis, by maturation of alveolar macrophages.

Molgramostim is a non-glycosylated recombinant human granulocyte macrophage colony stimulating factor (rhGM-CSF) produced by using recombinant DNA technology via a bacterial (E. coli) expression system. Molgramostim is formulated in a sterile nebulizer solution (molgramostim nebulizer solution) which is supplied in vials containing 300 µg of molgramostim in 1.2 mL solution and is administered by inhalation via an investigational eFlow Nebulizer System (PARI Pharma GmbH).

Results of a completed randomized, placebo-controlled clinical trial support the safety, tolerability, and efficacy of inhaled molgramostim nebulizer solution as a treatment for autoimmune PAP patients.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients must:

1. Be ≥18 years of age at the time of signing the informed consent.
2. Agree to use a highly effective form of contraception (see Section 3.5).
3. Have a positive serum anti-granulocyte macrophage colony-stimulating factor (GM CSF) autoantibody test result confirming aPAP.
4. Have a history of pulmonary alveolar proteinosis (PAP), based on examination of a lung biopsy, bronchoalveolar lavage (BAL) cytology, or a high-resolution computed tomogram (HRCT) of the chest.
5. Have at least one symptom of aPAP, including but not limited to dyspnea (at rest or with exertion), cough, or fatigue.
6. Be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
7. Be willing and able to comply with the visit schedule and treatment plan specified in the protocol, as judged by the physician.

Exclusion Criteria:

Eligible patients must not:

1. Have a diagnosis of hereditary or secondary PAP, or a metabolic disorder of surfactant production.
2. Require a whole lung lavage (WLL) at the time of screening (patient may be eligible 1 week post WLL).
3. Have received GM-CSF treatment within 1 month prior to the screening visit.
4. Have been treated with any investigational product within 5 half-lives or 3 months (whichever is longer) prior to the screening visit.
5. Have a history of allergic reactions to GM-CSF or any of the excipients in the nebulizer solution.
6. Be using significant (e.g., more than 10 mg/day systemic prednisolone) immunosuppression.
7. Have a history of severe and unexplained side effects during aerosol delivery of any medicinal product.
8. Have a history or current diagnosis of a myeloproliferative disease or leukemia.
9. Have any other medical condition which in the opinion of the physician would make the patient unsuitable for treatment with molgramostim nebulizer solution.
10. Be pregnant or breastfeeding, or planning to become pregnant during treatment with molgramostim nebulizer solution.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Los Angeles, California
  - University Florida Health, Gainesville, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UT Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Background] Bogunovic M, Ginhoux F, Helft J, Shang L, Hashimoto D, Greter M, Liu K, Jakubzick C, Ingersoll MA, Leboeuf M, Stanley ER, Nussenzweig M, Lira SA, Randolph GJ, Merad M. Origin of the lamina propria dendritic cell network. Immunity. 2009 Sep 18;31(3):513-25. doi: 10.1016/j.immuni.2009.08.010. Epub 2009 Sep 10. PMID 19733489
- [Background] Hamilton JA. Colony-stimulating factors in inflammation and autoimmunity. Nat Rev Immunol. 2008 Jul;8(7):533-44. doi: 10.1038/nri2356. PMID 18551128
- [Background] Inaba K, Inaba M, Romani N, Aya H, Deguchi M, Ikehara S, Muramatsu S, Steinman RM. Generation of large numbers of dendritic cells from mouse bone marrow cultures supplemented with granulocyte/macrophage colony-stimulating factor. J Exp Med. 1992 Dec 1;176(6):1693-702. doi: 10.1084/jem.176.6.1693. PMID 1460426
- [Background] Khan A, Agarwal R. Pulmonary alveolar proteinosis. Respir Care. 2011 Jul;56(7):1016-28. doi: 10.4187/respcare.01125. Epub 2011 Apr 15. PMID 21496372
- [Background] Kumar A, Abdelmalak B, Inoue Y, Culver DA. Pulmonary alveolar proteinosis in adults: pathophysiology and clinical approach. Lancet Respir Med. 2018 Jul;6(7):554-565. doi: 10.1016/S2213-2600(18)30043-2. Epub 2018 Feb 1. PMID 29397349
- [Background] McCarthy C, Avetisyan R, Carey BC, Chalk C, Trapnell BC. Prevalence and healthcare burden of pulmonary alveolar proteinosis. Orphanet J Rare Dis. 2018 Jul 31;13(1):129. doi: 10.1186/s13023-018-0846-y. PMID 30064481
- [Background] McCarthy C, Carey BC, Trapnell BC. Autoimmune Pulmonary Alveolar Proteinosis. Am J Respir Crit Care Med. 2022 May 1;205(9):1016-1035. doi: 10.1164/rccm.202112-2742SO. PMID 35227171
- [Background] Metcalf D. The molecular biology and functions of the granulocyte-macrophage colony-stimulating factors. Blood. 1986 Feb;67(2):257-67. PMID 3002522
- [Background] Park LS, Friend D, Gillis S, Urdal DL. Characterization of the cell surface receptor for human granulocyte/macrophage colony-stimulating factor. J Exp Med. 1986 Jul 1;164(1):251-62. doi: 10.1084/jem.164.1.251. PMID 3014035
- [Background] Trapnell BC, Carey BC, Uchida K, Suzuki T. Pulmonary alveolar proteinosis, a primary immunodeficiency of impaired GM-CSF stimulation of macrophages. Curr Opin Immunol. 2009 Oct;21(5):514-21. doi: 10.1016/j.coi.2009.09.004. Epub 2009 Sep 30. PMID 19796925
- [Background] Trapnell BC, Nakata K, Bonella F, Campo I, Griese M, Hamilton J, Wang T, Morgan C, Cottin V, McCarthy C. Pulmonary alveolar proteinosis. Nat Rev Dis Primers. 2019 Mar 7;5(1):16. doi: 10.1038/s41572-019-0066-3. PMID 30846703
- [Background] Trapnell BC, Inoue Y, Bonella F, Morgan C, Jouneau S, Bendstrup E, Campo I, Papiris SA, Yamaguchi E, Cetinkaya E, Ilkovich MM, Kramer MR, Veltkamp M, Kreuter M, Baba T, Ganslandt C, Tarnow I, Waterer G, Jouhikainen T; IMPALA Trial Investigators. Inhaled Molgramostim Therapy in Autoimmune Pulmonary Alveolar Proteinosis. N Engl J Med. 2020 Oct 22;383(17):1635-1644. doi: 10.1056/NEJMoa1913590. Epub 2020 Sep 7. PMID 32897035